CLINICAL TRIAL: NCT05810948
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Proof-of-Concept Study to Evaluate the Efficacy and Safety of Efgartigimod in Chinese Patients With Lupus Nephritis
Brief Title: A Study to Assess Effectiveness and Safety of Efgartigimod in Chinese Patients With Lupus Nephritis (ZL-1103-013)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2202
Record Dates: First submitted 2022-12-19; First posted 2023-04-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Lupus Nephritis
Keywords: Nephritis; Lupus Nephritis; Kidney Disease; Urologic Disease; Glomerulonephritis
MeSH Terms: conditions — Lupus Nephritis; Nephritis; Kidney Diseases; Urologic Diseases; Glomerulonephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- efgartigimod IV (Experimental): Patients receiving intravenous (IV) infusions of efgartigimod
  Interventions: Biological: efgartigimod IV
- Placebo (Placebo Comparator): Patients receiving intravenous (IV) infusions of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: efgartigimod IV — Intravenous (IV) infusion of efgartigimod
  Arms: efgartigimod IV
Other: Placebo — Intravenous (IV) infusion of placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of efgartigimod IV in Chinese patients with active lupus nephritis (LN). The study comprises an approximate 4-week screening period, a 24-week treatment period, and an 8-week follow- up period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years when signing the informed consent form (ICF)
* Capable of providing signed informed consent, and complying with protocol requirements
* Diagnosis of SLE according to the Systemic Lupus Erythematosus International Collaborating Clinic (SLICC) 2012 classification criteria
* Active, proliferative LN Class III or IV [excluding Class III (C), IV-S (C), and IV-G (C)], either with or without the presence of Class V using the 2003 International Society of Nephrology (ISN)/Renal Pathology Society (RPS) criteria, proven by kidney biopsy within 6 months before randomization and confirmed by the central biopsy reading group
* Require LN induction therapy (glucocorticoids and MMF/MPA) based on investigator's clinical judgment. Induction therapy may begin before screening but should be initiated within 60 days before randomization
* Agree to use contraceptives consistent with local regulations. Full inclusion criteria can be found in the protocol

Exclusion Criteria:

* Active or chronic infection requiring treatment
* Any evidence of central nervous system lupus (including but not limited to seizures, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis, or CNS vasculitis)
* Currently on renal dialysis or expected to require dialysis during study period
* Previous kidney transplantation or planned transplantation during study period
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before randomization. The following cancers are not exclusionary: basal cell or squamous cell skin cancer; carcinoma in situ of the cervix; carcinoma in situ of the breast; incidental histological finding of prostate cancer
* Heart failure due to Systemic Lupus Erythematodes, or any other severe cardiovascular involvement with safety concerns according to investigator's judgment
* Any other known autoimmune disease that would interfere with an accurate assessment of clinical symptoms of SLE/LN or put the participant at undue risk
* Previously failed treatment with MMF or any form of mycophenolate-based induction therapy, based on the investigator's opinion
* Use of complementary therapies, including Traditional Chinese Medicine, herbs, or procedure (eg, acupuncture) that can potentially interfere with the efficacy and safety of participants as assessed by the investigator
* SARS-CoV-2 antigen-based positive test at screening. The test is required regardless of whether the participant has been vaccinated
* Known hypersensitivity or contraindication to efgartigimod, any excipient of the IMP, or SoC medication used in the study
* In the opinion of the investigator, current or history of (ie, within 12 months of randomization) alcohol, drug, or medication abuse
* Pregnant or lactating females and those who intend to become pregnant during study participation
* Any conditions or circumstances that in the opinion of the investigator may make the participant unsuitable for the study

The full list of criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in urine protein creatinine ratio (UPCR) | up to 24 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving complete renal response (CRR) at week 24 | up to 24 weeks
Time to complete renal response (CRR) | up to 32 weeks
Proportion of participants achieving partial renal response at week 24 | up to 24 weeks
Time to partial renal response (PRR) | up to 24 weeks
Change from baseline to week 24 in estimated glomerular filtration rate (eGFR) | up to 24 weeks
Change from baseline to week 24 in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K score | up to 24 weeks
Change from baseline to week 24 in the dosage of glucocorticoids | up to 24 weeks
Treatment failure rate during treatment period | up to 24 weeks
Proportion of participants achieving modified complete renal response (mCRR) at week 24 | up to 24 weeks
Efgartigimod serum concentration-time profile | up to 32 weeks
Changes from baseline in levels of total IgG | up to 32 weeks
Incidence of ADA against efgartigimod | up to 32 weeks
Median changes in concentration from baseline over time in biomarkers (Anti-dsDNA, C3, C4 and CH50) | up to 32 weeks
  (all have the same measuring units)
Change from baseline to week 24 in EuroQoL 5-Dimension 5-Level (EQ-5D-5L) score | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Peking University Third Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Hunan Provincial People's Hospital, Changsha
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital,Sun Yat-sen University, Guanzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - First Affiliated Hospital of University of South China, Hengyang
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huainan
  - Jieyang People's Hospital, Jieyang
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Liu Zhou Works Hospital, Liuchow
  - Jiangxi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Huashan Hospital Fudan University, Shanghai
  - ShengJing Hospital of China Medical University, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijia Zhuang
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Shaanxi Provincial Hospital of Chinese Medicine, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided